CLINICAL TRIAL: NCT03386656
Title: Randomized, Placebo-controlled, Double-blind Trial to Evaluate the Efficacy and Safety of Topical Application of Tranexamic Acid for Saving Blood Losses in Patients Subjected to Prosthetic Knee Surgery
Brief Title: Efficacy and Safety of Topical Application of Tranexamic Acid for Saving Blood Losses in Patients Subjected to Prosthetic Knee Surgery
Acronym: TRA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación Pública Andaluza Progreso y Salud (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FPS-TRA-2017-02
Record Dates: First submitted 2017-06-26; First posted 2017-12-29 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; Tranexamic acid
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Amchafibrin (Experimental): Estimated total blood loss, measured using the formula described by Nadler. A difference in estimated blood loss greater than or equal to 245 ml will be considered clinically relevant.
  Interventions: Drug: Amchafibrin
- Saline Solution 0,9%. (Placebo Comparator): Comparator of tranexamic acid
  Interventions: Other: Saline Solution

INTERVENTIONS:
Drug: Amchafibrin — Tranexamic acid (Amchafibrin) exerts an antihemorrhagic activity by inhibiting the fibrinolytic properties of plasmin.
  Arms: Amchafibrin
Other: Saline Solution — Placebo
  Other Names: Placebo
  Arms: Saline Solution 0,9%.

SUMMARY:
To compare the efficacy and safety of topical tranexamic acid versus placebo in patients diagnosed with severe knee osteoarthritis who will undergo prosthetic knee surgery in terms of saving blood loss (estimated blood loss, decreased hemoglobin and Decrease in hematocrit).

DETAILED DESCRIPTION:
Tranexamic acid (Amchafibrin) exerts an antihemorrhagic activity by inhibiting the fibrinolytic properties of plasmin. Tranexamic acid binds to plasminogen when it is transformed into plasmin. The activity of the tranexamic acid-plasmin complex on fibrin activity is less than the activity of free plasmin alone.

There are two methods of presentation: one, as an injectable solution; Two as a clear, colorless aqueous solution.

Tranexamic acid in Spain is approved for use in the prevention and treatment of bleeding due to general fibrinolysis. As for its specific indications the investigators find that it is used for the treatment of metrorrhagia, menorrhagia, gastrointestinal hemorrhage, urinary hemorrhagic disorders after prostate surgery, surgery of ears, nose, throat, gynecological, thoracic, abdominal or cardiovascular or to counter associated hemorrhages To the administration of a fibrinolytic drug.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, in the age group: ≥18 and ≤80 years.
* Patients diagnosed with confirmation of severe knee osteoarthritis according to Kellgren criteria (equal or greater than 2) and EVA greater than 7, who will be subjected to knee arthroplasty surgery.
* Patients signing informed consent, agreeing to participate in the study.

Exclusion Criteria:

* Patients with concomitant cardiac disease: unstable angina pectoris, acute myocardial infarction, atrial fibrillation, flutter, history of sudden death, severe valve insufficiency.
* Patients with concomitant previous thromboembolic disease: Deep venous thrombosis, pulmonary thromboembolism, thrombotic arterial embolism, Ischemic Vascular Cerebral Stroke, fibrinolytic diseases after consumption coagulopathy.
* Hypersensitivity to tranexamic acid.
* Severe systemic disease: cardio-pulmonary, neurological, renal, infectious or any other type that may impede the development of the study or evaluation of the results.
* History of seizures.
* Patients with severe mental disorder (psychotic disorder, risk of autolysis, manic episode), dependence on toxic substances and / or some physical or psychological limitation to answer.
* Patients receiving oral anticoagulants.
* Patients in litigation for disability claim related or not with the disease.
* Patients who cannot make the necessary visits to carry out the study.
* Patients who refuse to participate or sign informed consent.
* Pregnant and lactating patient's period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-08 (Actual)

PRIMARY OUTCOMES:
Saving blood loss in knee surgery | 24 hours post-intervention
  Total blood loss greater than 245 ml

SECONDARY OUTCOMES:
Time post-intervention of functional recovery in study subjects | Four weeks post-discharger
Length of hospital stay in study subjects | Four weeks post-discharger

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Puerta del Mar, Cadiz, Spain

IPD SHARING:
Plan to Share IPD: Undecided